CLINICAL TRIAL: NCT06115694
Title: Comparison of Video Laryngoscopy With Rigid Stylet vs Video Laryngoscopy With the TCI Articulating Introducer for Endotracheal Intubation in Simulated Difficult Airways:A Prospective Randomized Controlled Multicenter Study
Brief Title: Comparison of Video Laryngoscopy With Rigid Stylet vs Video Laryngoscopy With the TCI Articulating Introducer for Endotracheal Intubation in Simulated Difficult Airways
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GWang025
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Intubation; Difficult or Failed
Keywords: TCI Articulating Introducer; Endotracheal cannula; Simulated difficult airway

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group：TCI Articulating Introducer (Active Comparator): Tracheal intubation was performed using a TCI core under a visual laryngoscope
  Interventions: Device: TCI Articulating Introducer
- Control group：GlideRite® Rigid Stylet (Placebo Comparator): Tracheal intubation was performed under a visual laryngoscope using a common tube core
  Interventions: Device: GlideRite® Rigid Stylet

INTERVENTIONS:
Device: TCI Articulating Introducer — use
  Arms: Experimental group：TCI Articulating Introducer
Device: GlideRite® Rigid Stylet — use
  Arms: Control group：GlideRite® Rigid Stylet

SUMMARY:
Purpose:

To compare the efficacy and safety of TCI tube core and ordinary tube core assisted tracheal intubation in simulating difficult airway under visual laryngoscope, and to provide reference for clinical application

DETAILED DESCRIPTION:
Endotracheal intubation plays an important role in contemporary clinical anesthesia. Direct laryngoscope intubation is the traditional intubation method in anesthesia and emergency medical work. However, due to the constraints of the operator's technical level, the abnormal airway structure and the condition of patients, about 1.5% ~ 8.5% of the cases of intubation difficulties occur. It's even impossible to intubate. Failure of intubation can lead to major complications, including brain damage and death. When a tracheal intubation cannot be placed on the first two attempts, the intubation is classified as difficult, and repeated routine tracheal intubation may lead to morbidity in the patient, and the incidence of airway related complications increases significantly with the number of tracheal intubations. Difficult intubation accounted for 4% of operating room intubation and 10% of intubation outside the operating room. For patients with high glottis and short epiglottis, although the glottis can be seen, intubation is difficult to place. The effectiveness and safety of TCI tube assisted intubation under visual laryngoscope and ordinary tube tube assisted intubation in simulated difficult airway were compared to provide reference for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥18 years of age or non-pregnant women;
2. For elective gynecological surgery or upper abdominal surgery under general anesthesia by oral tracheal intubation, the operation position was supine and the operation time was less than 3 hours;
3. Subject's American Society of Anesthesiologists physical status is I-III
4. Subjects who could understand the purpose of the trial, voluntarily participated and signed the informed consent form, and were willing to accept the designated follow-up.

Exclusion Criteria:

1. any cerebrovascular accident, such as stroke, transient ischemic attack (TIA), etc. occurred within 3 months;
2. patients with unstable angina pectoris or myocardial infarction within 3 months;
3. laryngeal mass, obstruction, maxillofacial fracture or deformity;
4. Full stomach, high intra-abdominal pressure, habitual vomiting, gastroesophageal reflux disease;
5. pharyngeal infection, hematoma, abscess, tonsil enlargement;
6. Upper respiratory tract infection within one month, fever, cough, runny nose, nasal congestion, etc.;
7. history of chronic airway inflammation, airway hyperresponsiveness or asthma;
8. diabetic patients with severe diabetic complications (diabetic ketoacidosis, hyperosmolar coma, various infections, macroangiopathy, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot, etc.);
9. severe complications of hypertension, such as arterial dissection, renal failure, cerebral hemorrhage, etc.;
10. reoperation within 3 months;
11. patients with contraindications or allergies to intraoperative drugs;
12. patients enrolled in other studies within 30 days;
13. poor adherence or the investigator's opinion that the patient was not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The success of intubation for the first time | 1 day of surgery
  To compare the success rate of first intubation in simulated difficult airway with TCI tube assisted by visual laryngoscope and ordinary tube.

SECONDARY OUTCOMES:
Overall success rate of intubation | 1 day of surgery
  Overall success rate of tracheal intubation assisted by TCI and conventional tube cores under video laryngoscope in all included patients
Whether it is necessary to rotate the tracheal tube through the glottis | 1 day of surgery
  Whether it is necessary to rotate during tracheal intubation to successfully enter the airway through the glottis
Throat complications | 24 hours after surgery
  Whether the following conditions will occur after operation: oral mucosal injury: tracheal tube stained with blood or secretion with blood when extubation; Sore throat: patients complained of throat discomfort, manifested as slurred speech, foreign body sensation, cough, etc. Loose teeth; Difficulty speaking; Patients were followed up for 24 hours after surgery to see whether they still had dysphagia, nausea, vomiting, and cough.

IPD SHARING:
Plan to Share IPD: No